CLINICAL TRIAL: NCT04302480
Title: A Brief Intervention Programme on Alternative Smoking Products
Brief Title: A Brief Intervention Programme on ASP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Daniel Sai-Yin Ho, Principle investigator and associate professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: coshdrama2020
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Alternative Smoking Products
MeSH Terms: interventions — aspartyl-aspartic acid; SSB protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternative smoking products (ASP) (Experimental)
  Interventions: Other: Worksheets for ASP; Other: E-messages for ASP
- Sugar-sweetened beverages (SSB) (Active Comparator)
  Interventions: Other: Worksheets for SSB; Other: E-messages for SSB

INTERVENTIONS:
Other: Worksheets for ASP — The ASP intervention will cover the harms and misleading marketing strategies of ASPs and other related information.
  Arms: Alternative smoking products (ASP)
Other: Worksheets for SSB — The SSB intervention will cover the general information on SSBs, such as the sugar content of SSBs, nutrition labels and the harms of SSBs.
  Arms: Sugar-sweetened beverages (SSB)
Other: E-messages for ASP — In the subsequent month after the main intervention, students in the ASP group will receive 4-6 e-messages on ASPs, after which students will be invited to complete a 1-month follow-up assessment.
  Arms: Alternative smoking products (ASP)
Other: E-messages for SSB — In the subsequent month after the main intervention, students in the SSB group will receive 4-6 e-messages on SSBs, after which students will be invited to complete a 1-month follow-up assessment.
  Arms: Sugar-sweetened beverages (SSB)

SUMMARY:
The brief intervention comprises a 4-page worksheet used in the classroom (main intervention) and subsequent weekly e-messages through WhatsApp (booster intervention). The worksheets for both groups will be printed in colour, and mainly contain pictures and simple texts. Students will be asked to provide smartphone numbers of themselves and their parents for receiving the booster interventions. After sending 4-6 e-messages in 4 weeks, students will complete a 1-month follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Parents and children should understand Chinese.
* Parents' consent to their children's participation.

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-05-18 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Knowledge on the harms and misleading marketing strategies of ASPs | Immediately after intervention
  Students will report their opinions towards 5 statements:
  1. Children who use e-cigarettes are more likely to smoke cigarettes in the future;
  2. Hazards of secondhand smoke of e-cigarettes and heated tobacco products are slight;
  3. Nicotine content in heated tobacco products is lower than in the cigarettes, which is more difficult to get addicted;
  4. There are a variety of carcinogens in the heated tobacco products;
  5. Tobacco industries do everything they can to get young people to use tobacco products.
  All the statements have 5 options from definitely no to definitely yes. The options will be recoded into 0-4 or 4-0, as appropriate, with higher scores indicating knowing more about the harms and misleading marketing strategies of ASPs.
Attitudes towards ASPs | Immediately after intervention
  Students will report their opinions towards 2 questions:
  1. Do you think the usage of e-cigarettes and heated tobacco products will harm your health?
     There will be 11 options from definitely no harm to definitely harm.
  2. Do you accept the primary students use e-cigarettes and heated tobacco products?
  There will be 11 options from definitely unacceptable to definitely acceptable.

SECONDARY OUTCOMES:
Intention to use ASPs | Immediately after intervention
  If one of your good friends offers you an e-cigarette or heated tobacco product, ask you to have a few puffs, and no one will know about this as no more smoking in the future. Will you use them?
  There will be 11 options from definitely no to definitely yes.
Knowledge on the harms and misleading marketing strategies of ASPs | 1-month follow-up
  Students will report their opinions towards 5 statements:
  1. Hazards of e-cigarettes are slight, can only cause minor health problems;
  2. Reliable evidence shows that e-cigarettes can help quit smoking cigarettes;
  3. Heated tobacco products contain tar, can cause a variety of cancers;
  4. Heated tobacco products are harm reduction products, which is less harmful than cigarettes;
  5. Tobacco industries conceal the harms of tobacco products for commercial gain.
  All the statements have 5 options from definitely no to definitely yes. The options will be recoded into 0-4 or 4-0, as appropriate, with higher scores indicating knowing more about the harms and misleading marketing strategies of ASPs.
Attitudes towards ASPs | 1-month follow-up
  Students will report their opinions towards 2 questions:
  1. Do you think the usage of e-cigarettes and heated tobacco products will harm your health?
     There will be 11 options from definitely no harm to definitely harm.
  2. Do you accept the primary students use e-cigarettes and heated tobacco products?
  There will be 11 options from definitely unacceptable to definitely acceptable.
Intention to use ASPs | 1-month follow-up
  If one of your good friends offers you an e-cigarette or heated tobacco product, ask you to have a few puffs, and no one will know about this as no more smoking in the future. Will you use them?
  There will be 11 options from definitely no to definitely yes.

CONTACTS AND LOCATIONS:
Overall Officials: Sai Yin Ho, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Local primary schools, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No